CLINICAL TRIAL: NCT06598657
Title: Effects of Talocrural Joint Mobilization With Movement in Spastic Cerebral Palsy Patients
Brief Title: Talocrural Mobilization With Movement in Spastic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01877 Maimoona Mubarik
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Spastic Cerebral Palsy (sCP)
Keywords: Talocrural joint; Mobilization with Movement; Spasticity cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with Movement MWM of Talocrural joint + Conventional PT (Active Comparator)
  Interventions: Other: Mobilization with Movement MWM
- Conventional PT (Other)
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Mobilization with Movement MWM — Mobilization with Movement MWM of Talocrural joint in non-weight bearing position to improve Dorsiflexion Range of Motion (3 sets of 6 repetitions were applied, with a 1-minute break between sets/3 times a week) and conventional therapy which includes stretching, strengthening, balance training exercise.
  Arms: Mobilization with Movement MWM of Talocrural joint + Conventional PT
Other: Conventional Treatment — * Stretches of Hamstrings, Gastrocnemius, Soleus and hip adductors with duration of 20 sec hold/ 5 reps and Frequency: 3 times/week. Stretches will be performed passively
  * Strengthening exercises of Quadriceps and abdominal muscles three times a week.
  * Static balance exercises including single leg balance, tandem stance, weight shifting with Duration: 10 sec hold/ 5 reps Frequency: 3 times/week
  Arms: Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to find the effect of Mulligan's Mobilization with Movement of Talocrural joint in Cerebral Palsy Patients having spasticity on improving Ankle Range of Motion, improving balance and its effect on Gait speed.

DETAILED DESCRIPTION:
Cerebral palsy is a neurodevelopmental disorder involving abnormalities in muscle tone and motor function due to damaged cerebral tissue in development. It is a nonprogressive upper motor neuron lesion characterized by abnormal tone, posture, balance and movement and clinically classified based on the predominant motor syndrome. In spastic CP, there is significant weakness that contributes to abnormal posture and movement. This is also accompanied by decreased muscle endurance and loss of selective motor control (SMC). Spastic diplegia is a very common form of CP, with a wide range of ambulatory outcomes, and is most frequently accompanied by ankle spasticity. Abnormalities, such as excessive plantar flexion of the ankle, leads to individuals with CP have in both static and dynamic balance.

Joint mobilization has not only the mechanical effect of disrupting the contracture by direct movement of the joint area, but also stimulates mechanoreceptor activation when stretching occurs in the capsule and ankle ligaments.

The Mulligan Mobilization with movement (MWM) is a physical therapy technique that combines joint mobilization techniques with active movement. It aims to improve joint range of motion, reduce stiffness, and enhance functional mobility, is expected to produce an instantaneous improvement in the patient's abilities by simultaneous applying of pain-free accessory glides.

This study will contribute in describing long lasting effects of Mobilization With Movement, with multiple assessments, on ankle range of motion, balance, and gait speed, and to check whether the amount of regaining is similar between patients undergoing MWM with conventional therapy and those with conventional therapy alone

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age group 8-18 years
* Diagnosis of spastic Cerebral Palsy
* CP to follow verbal directions
* Modified Ashworth Scale score of '1' or '1+'
* Function classification system (GMFCS) level I or II ability to walk
* 10 m or more independently

Exclusion Criteria:

* visual, hearing disorders
* verbal and cognitive disorders (unable to comprehend commands)
* recent lower extremity surgery
* botulinum toxin injection

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go | 4 weeks
  In the TUG test, a child begins in a seated position on a chair or other designated surface. They are instructed to stand up, walk a specific distance (usually three meters or ten feet), turn around, and return to the seated position. The time taken to complete the task is recorded. Evaluation is made by comparing pre and post-intervention. To assess mobility of patient.
10 m WALK TEST | 4 weeks
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility and gait. Stopwatch is used and the total time taken to ambulate 6 meters is recorded. Timing starts when the toes pass the 2-meter mark. Timing stops when the toes pass the 8-meter mark. The 6m is then divided by the total time taken (in seconds) to completed. The total time is recorded in m/s
Goniometer | 4 weeks
  It is an instrument that measures the available range of motion at a joint.
Modified Ashworth Scale (MAS) | 4 weeks
  Modified Ashworth Scale (MAS) is used to assess spasticity. Different grades from 0 to 4 are used to access increased tone and spasticity. With 0 referring to "No increase in tone" and 4 refers to "Affected part rigid in flexion/extension" The measurements are recorded at baseline, during treatment and after treatment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- PAF School for Persons With special Needs PNS, Islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No